CLINICAL TRIAL: NCT07016165
Title: Ciprofloxacin Versus Ceftazidime as Empirical Therapy of High-Risk Neutropenic Fever in Children With Hematologic Malignancies : A Randomized Controlled Trial
Brief Title: Ciprofloxacin vs Ceftazidime for Empirical Treatment of High-Risk Neutropenic Fever in Children With Hematologic Malignancies
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Bambang Ardianto, Principal Investigator, Head of Pediatric Hematolo-Oncology Divison, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KE/FK/0517/EC/2025
Record Dates: First submitted 2025-05-30; First posted 2025-06-11 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Neutropenic Fever; Acute Lymphoblastic Leukemia; Acute Myeloblastic Leukemia; Non Hodgkin Lymphoma
Keywords: ciprofloxacin; ceftazidime; neutropenic fever; Acute Lymphoblastic Leukemia; Acute Myeloblastic Leukemia; Non Hodgkin Lymphoma
MeSH Terms: conditions — Febrile Neutropenia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin | interventions — Ceftazidime; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Standard therapy IV ciprofloxacin 10 mg/kgBW/12 hours
  Interventions: Drug: Ciprofloxacin
- Group B (Experimental): IV ceftazidime 150 mg/kgBW/24 hours divided into 3 doses
  Interventions: Drug: Ceftazidime

INTERVENTIONS:
Drug: Ceftazidime — Ceftazidime 150 mg/kgBW/24 hours divided into 3 doses.
  Arms: Group B
Drug: Ciprofloxacin — Ciprofloxacin 10 mg/kgBW/12 hours
  Arms: Group A

SUMMARY:
This clinical trial will compare use of ciprofloxacin and ceftazidime work in treating high-risk fever in children with hematological malignancies

1. Does ceftazidime work better than ciprofloxacin as a first-choice antibiotic for children with hematological malignancies who have high-risk fever from low neutrophil count?
2. Are there any specific factors that affect how children with hematological malignancies respond to ciprofloxacin or ceftazidime when treating high-risk fever?

Participants in this study are children with hematological malignancies who have a high risk of fever due to low neutrophil count. Children, aged 0 to 18 years old, will be hospitalized between June and December 2025 at Sardjito General Hospital

The study will involve:

* Collecting patient history, conducting physical exams, and performing supporting tests.
* Randomly assigning participants into two groups: one group will receive the standard treatment with intravenous ciprofloxacin, while the other group will receive the intervention treatment with intravenous ceftazidime.
* Both groups will be monitored for various outcomes, including the length of fever, length of low white blood cell count, length of hospital stay, length of antibiotic use, any changes in antibiotics, and mortality.

DETAILED DESCRIPTION:
Furthermore, this clinical trial aims to:

1. Compare the efficacy of empirical antibiotic administration of Ciprofloxacin and Ceftazidime in pediatric malignancy patients with high-risk neutropenic fever.
2. Analyze the differences in clinical effectiveness between ceftazidime and ciprofloxacin antibiotics based on the duration of fever, duration of neutropenia, duration of hospitalization in high-risk neutropenic fever in children with hematological malignancies.
3. Compare the mortality of pediatric patients with high-risk neutropenic fever due to hematological malignancies who received empirical antibiotic therapy of ceftazidime and ciprofloxacin.
4. Compare antibiotic escalation decisions in pediatric patients with high-risk neutropenic fever due to hematological malignancies who received empirical antibiotic therapy of ceftazidime and ciprofloxacin.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0 to 18 years with hematological malignancies.
* Children with high-risk neutropenic fever, namely children with blood malignancies induction phase ALL, consolidation phase ALL, reinduction phase ALL, relapse ALL; meningeal ALL, AML, and NHL, diagnosed by a competent pediatrician on duty.
* Consent from parents to be included in the study.

Exclusion Criteria:

* Children with malignancies but accompanied by comorbidities (HIV infection, septic shock).
* Allergy to ciproloxacin or ceftazidime.
* Fever associated with blood transfusion reactions.
* Receiving other antibiotics since 72 hours before being included in the study, except for cotrimoxazole prophylaxis for the prevention of Pneumocystis carinii pneumonia, and ciproloxacin prophylaxis in AML.
* Children with blood malignancies who have impaired renal function (serum creatinine ≥ 1.5 times the upper normal limit) and impaired liver function (SGPT > 5 times the upper normal limit).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of fever | from first administration of Ciprofloxacin or Ceftazidime to 48 hours fever free
  Duration of fever since receiving the first antibiotic, based on the temperature graph available in the electronic medical record
Duration of Neutropenia | From first antibiotic administration to 48 hours after administration
  The length of time the subject experiences neutropenia, absolute neutrophil count is <500

SECONDARY OUTCOMES:
Duration of hospitalization | From first administration of Ciprofloxacin or Ceftazidime to hospital discharge
  The duration from the date of subject recruitment to the date of hospital discharge, as recorded in the electronic medical record.
Duration of antibiotic use | days from first administration to the last intravenous antibiotic administration
  days of antibiotic use from the first administration to the last intravenous antibiotic administration
Antibiotic escalation decisions | From first administration of Ciprofloxacin or Ceftazidime to 48 hours after administration
  Clinician decisions in escalating empirical antibiotics to second-line antibiotics
Mortality | from first administration of ciprofloxacin or ceftazidime to 30 days after recruitment
  Mortality of subject in admission is proven by a death certificate

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP dr Sardjito, Sleman, DI Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be considered after completion of ongoing analyses

REFERENCES:
- [Background] Corapcioglu F, Sarper N. Cefepime versus ceftazidime + amikacin as empirical therapy for febrile neutropenia in children with cancer: a prospective randomized trial of the treatment efficacy and cost. Pediatr Hematol Oncol. 2005 Jan-Feb;22(1):59-70. doi: 10.1080/08880010590896297. PMID 15770833
- [Background] Kamonrattana R, Sathitsamitphong L, Choeyprasert W, Charoenkwan P, Natesirinilkul R, Fanhchaksai K. A Randomized, Open-Labeled, Prospective Controlled Study to Assess the Efficacy of Frontline Empirical Intravenous Piperacillin/Tazobactam Monotherapy in Comparison with Ceftazidime Plus Amikacin for Febrile Neutropenia in Pediatric Oncology Patients. Asian Pac J Cancer Prev. 2019 Sep 1;20(9):2733-2737. doi: 10.31557/APJCP.2019.20.9.2733. PMID 31554370
- [Background] Yasuda T, Suzuki R, Ishikawa Y, Terakura S, Inamoto Y, Yanada M, Nagai H, Ozawa Y, Ozeki K, Atsuta Y, Emi N, Naoe T. Randomized controlled trial comparing ciprofloxacin and cefepime in febrile neutropenic patients with hematological malignancies. Int J Infect Dis. 2013 Jun;17(6):e385-90. doi: 10.1016/j.ijid.2012.12.005. Epub 2013 Jan 11. PMID 23317527